CLINICAL TRIAL: NCT01384383
Title: A Phase 2 Randomized, Open-Label, Exploratory Trial of GS-5885, GS-9451 With Peginterferon Alfa 2a and Ribavirin (RBV) in Treatment-Naïve Subjects With Chronic Genotype 1 Hepatitis C Virus Infection and IL28B CC Genotype
Brief Title: GS-5885, GS-9451 With Peginterferon Alfa 2a (PEG) and Ribavirin in Treatment-Naïve Subjects With Chronic Genotype 1 Hep C Virus Infection and IL28B CC Genotype
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-248-0121
Record Dates: First submitted 2011-06-22; First posted 2011-06-29 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; IL28B CC Genotype; Treatment naive; Peginterferon α-2a (PEG); Genotype 1a/b; GS 9451; GS 5885; Ribavirin (RBV); HCV NS5A inhibitor; HCV NS3 protease inhibitor
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ledipasvir; GS-9451

ARMS (2):
- Arm 1 (Experimental): Response-Guided Therapy with GS-5885 30 mg plus GS-9451 200 mg, plus PEG and RBV for 6 or 12 weeks.
  Interventions: Drug: GS-5885; Drug: GS-9451; Drug: RBV; Drug: PEG
- Arm 2 (Experimental): Response-Guided Therapy with PEG and RBV for 24 weeks.
  Interventions: Drug: RBV; Drug: PEG

INTERVENTIONS:
Drug: GS-5885 — GS-5885 30 mg tablet administered orally once daily
  Arms: Arm 1
Drug: GS-9451 — GS-9451 200 mg tablet administered orally once daily
  Arms: Arm 1
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)
Drug: PEG — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection

SUMMARY:
This is a Phase 2, randomized, open-label exploratory study that will examine the antiviral efficacy, safety, and tolerability of Response guided treatment (RGT) with GS-5885 + GS-9451 + PEG/RBV (6 or 12 weeks), or Peginterferon Alfa 2a (PEG)/Ribavirin (RBV)alone (24 weeks) in treatment naïve subjects with chronic Hep C (HCV) infection with genotype (GT) 1 and IL28B CC genotype.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-70 years of age
* Chronic HCV infection
* Subjects must have liver biopsy results (≤ 3 years prior to screening) indicating the absence of cirrhosis. Alternatively a non-invasive alternative to liver biopsy (such as FibroTest, FibroScan, or Acoustic Radiation Force Impulse imaging) within 6 months of Screening in countries where allowed
* Monoinfection with HCV genotype 1a or 1b
* HCV RNA > 10^4 IU/mL at Screening
* IL28B CC genotype
* HCV treatment naïve
* Candidate for PEG/RBV therapy
* Body mass index (BMI) between 18 and 36 kg/m2
* Creatinine clearance >= 50 mL/min
* Agree to use two forms of highly effective contraception methods for the duration of the study and for 7 months after the last dose study medication. Females of childbearing potential must have negative pregnancy test at Screening and Baseline

Exclusion Criteria:

* Exceed defined thresholds for key laboratory parameters at Screening
* Diagnosis of autoimmune disease, decompensated liver disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease (COPD), HIV, hepatitis B virus (HBV), hepatocellular carcinoma or other malignancy (with exception of certain skin cancers), hemoglobinopathy, retinal disease, or are immunosuppressed
* Subjects with current use of amphetamines, cocaine, opiates (e.g., morphine, heroin), or ongoing alcohol abuse are excluded. Subjects on stable methadone maintenance treatment for at least 6 months prior to Screening may be included into the study
* Use of prohibited concomitant medications two weeks prior to baseline through the end of treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | 30 , 36 or 48 weeks
  Sustained virologic response (SVR, defined as plasma HCV RNA < lower limit of quantification [LLoQ] at 24 weeks after treatment cessation) following treatment with GS-5885 + GS-9451 + PEG/RBV for 6 or 12 weeks, or PEG/RBV for 24 weeks in IL28B CC subjects.

SECONDARY OUTCOMES:
Safety and tolerability of therapy | Up to 48 weeks
  Safety and tolerability of the therapy is measured by frequency of laboratory abnormalities , reported adverse events and discontinuations due to adverse events.
Virologic response | Weeks 2, 4, 6, 8, 10, and 12
  Virologic response at Weeks 2, 4, 6, 8, 10, and 12 (depending on treatment arm) as measured by the rates of HCV RNA < LLoQ and viral breakthrough and relapse
Compare SVR | Weeks 30 and 36
  Compare SVR following treatment with GS-5885 + GS-9451 + PEG/RBV for 6 weeks versus 12 weeks.
Viral resistance | Up to 96 Weeks
  Characterize viral resistance to GS-5885 and GS-9451 when administered in combination with PEG/RBV

CONTACTS AND LOCATIONS:
Locations (54):
- United States (25):
  - Axis Clinical Trials, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - V.A. Greater Los Angeles Healthcare System, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Research and Education, Inc., San Diego, California
  - San Jose Gastroenterology, San Jose, California
  - Stanford University, Stanford, California
  - South Denver Gastroenterology, Englewood, Colorado
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Commonwealth Clinical Studies, LLC, Brockton, Massachusetts
  - Impact Clinical Trials, Las Vegas, Nevada
  - North Shore University Hospital, Great Neck, New York
  - Weill Cornell College of Medicine, New York, New York
  - Westchester Medical Center, Yonkers, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - The North Texas Research Institute, Arlington, Texas
  - Research Specialists of Texas, Houston, Texas
  - University of Utah Pediatric Pulmonology, Salt Lake City, Utah
  - Metropolitan Liver Diseases Center, Fairfax, Virginia
  - Liver Institute of Virginia, Bon Secours Health System, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Harborview Medical Center, Seattle, Washington
- Australia (20):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Saint Vincents Hospital, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane Hospital Research Foundation, Herston, Queensland
  - Greenslopes Private Hospital, Woolloongabba, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - St. Vincent's Hospital, Sydney Ltd., Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria
  - Austin Health, Department of Hepatology, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - LAIR Centre, Vancouver, British Columbia
  - GIRI GI Research Institute, Vancouver, British Columbia
  - University of Manitoba, John Buhler Research Centre, Winnipeg, Manitoba
  - London Health Sciences, London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- New Zealand (2):
  - Auckland Hospital, Aukland
  - Waikato Hospital, Hamilton